CLINICAL TRIAL: NCT06599541
Title: Efficacy of Hypopressive Exercises Versus Pilates in Women with Abdominal Diastasis in the Postpartum Period: a Randomized Controlled Trial
Acronym: AD-HE-PI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Adrián Rosales Torrejón, Principal Investigator, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Abdominal diastasis
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Abdominal Diastasis
Keywords: Hypopressive Exercise; Pilates; Abdominal Diastasis; Postpartum
MeSH Terms: interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HE group (Experimental): Participants with AD who are going to perform hypopressive exercises
  Interventions: Behavioral: Hypopressive Exercise
- Pilates group (Experimental): Participants with AD who are going to perform pilates exercises.
  Interventions: Behavioral: Pilates Exercise

INTERVENTIONS:
Behavioral: Hypopressive Exercise — A hypopressive exercise program will be carry out.
  Arms: HE group
Behavioral: Pilates Exercise — A pilates exercise program will be carry out.
  Arms: Pilates group

SUMMARY:
The aim of this study is to compare the effects of two exercise programs in women with abdominal diastasis (AD) during the postpartum. One group will receive hypopressive exercises (HE) and the other will receive pilates exercise. The hypothesis of this study is that the execution of both protocols will offer benefits in the ultrasound values of the AD and in the data collected on the quality of life in the short term and 12 weeks after its completion.

DETAILED DESCRIPTION:
Objective: To compare the efficacy of hypopressive exercises (HE) versus pilates exercise in women with abdominal diastasis (AD) during the postpartum, and to know the effects of each of the exercises independently.

Design: Single-blind randomized controlled trial.

Setting: Faculty of Physical Therapy of Alcalá de Henares (UAH).

Participants: Primiparous women with DA who have vaginal delivery and are in the 3 months postpartum (N=40).

Interventions: Participants will be randomly assigned to perform either a HE program focused on freediving work (n=20) or a pilates program focused on exhalation (n=20). The intervention will consist of 3 weekly sessions lasting 30 minutes over 12 weeks, where they will receive a weekly face-to-face and group session and two home sessions.

Main outcome measures: The primary outcome will be measurement of the distance between rectus abdominis through ultrasound to be assessed at baseline, immediately after the intervention and 12 weeks later. The secondary outcome measure will correspond to the measurement of quality of life using the SF-36 Health Questionnaire. It will be collected through masked evaluations by 2 physiotherapists at baseline, at the end of the intervention and at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women over 18 years of age who are within 3 months postpartum.
* AD with values >2.5 cm in any of the following reference points: 2 cm supraumbilical or 2 cm infraumbilical.
* Vaginal birth.

Exclusion Criteria:

* Abdominal or umbilical hernia.
* Previous abdominal surgery.
* Be receiving any other treatment for your AD

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Distance between rectus abdominis. | The measurements will be collected at baseline, immediately after the treatment and 12 weeks after the end of treatment.
  The distance between both muscle bellies of the rectus abdominis will be measured with an ultrasound (linear probe). It will be measured at two reference points: 2 cm supraumbilical and 2 cm infraumbilical.

SECONDARY OUTCOMES:
Quality of life | The scale will be passed at baseline, immediately after the treatment and 12 weeks after the end of treatment.
  The SF-36 consists of a health questionnaire composed of 36 items for the characterization of a person´s health. The total score ranges between 0 and 100 points. A higher score reflects more optimal health.

CONTACTS AND LOCATIONS:
Overall Officials: Adrián Rosales Torrejón, MSc, Principal Investigator — University of Alcala; Ana Serrano Imedio, PdH, Study Director — University of Alcala
Locations (1):
- Campus Científico Tecnológico UAH. Av. de León, 3A, Fuenlabrada, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gluppe S, Engh ME, Bo K. What is the evidence for abdominal and pelvic floor muscle training to treat diastasis recti abdominis postpartum? A systematic review with meta-analysis. Braz J Phys Ther. 2021 Nov-Dec;25(6):664-675. doi: 10.1016/j.bjpt.2021.06.006. Epub 2021 Jul 21. PMID 34391661
- [Background] Liaw LJ, Hsu MJ, Liao CF, Liu MF, Hsu AT. The relationships between inter-recti distance measured by ultrasound imaging and abdominal muscle function in postpartum women: a 6-month follow-up study. J Orthop Sports Phys Ther. 2011 Jun;41(6):435-43. doi: 10.2519/jospt.2011.3507. Epub 2011 Feb 2. PMID 21289454
- [Background] Mazzarino M, Kerr D, Wajswelner H, Morris ME. Pilates Method for Women's Health: Systematic Review of Randomized Controlled Trials. Arch Phys Med Rehabil. 2015 Dec;96(12):2231-42. doi: 10.1016/j.apmr.2015.04.005. Epub 2015 Apr 23. PMID 25912668
- [Background] Gluppe SL, Hilde G, Tennfjord MK, Engh ME, Bo K. Effect of a Postpartum Training Program on the Prevalence of Diastasis Recti Abdominis in Postpartum Primiparous Women: A Randomized Controlled Trial. Phys Ther. 2018 Apr 1;98(4):260-268. doi: 10.1093/ptj/pzy008. PMID 29351646
- [Background] Mota P, Pascoal AG, Carita AI, Bo K. The Immediate Effects on Inter-rectus Distance of Abdominal Crunch and Drawing-in Exercises During Pregnancy and the Postpartum Period. J Orthop Sports Phys Ther. 2015 Oct;45(10):781-8. doi: 10.2519/jospt.2015.5459. Epub 2015 Aug 24. PMID 26304639
- [Background] Vicente-Campos D, Sanchez-Jorge S, Terron-Manrique P, Guisard M, Collin M, Castano B, Rodriguez-Sanz D, Becerro-de-Bengoa-Vallejo R, Chicharro JL, Calvo-Lobo C. The Main Role of Diaphragm Muscle as a Mechanism of Hypopressive Abdominal Gymnastics to Improve Non-Specific Chronic Low Back Pain: A Randomized Controlled Trial. J Clin Med. 2021 Oct 27;10(21):4983. doi: 10.3390/jcm10214983. PMID 34768502
- [Background] Ramirez-Jimenez M, Alburquerque-Sendin F, Garrido-Castro JL, Rodrigues-de-Souza D. Effects of hypopressive exercises on post-partum abdominal diastasis, trunk circumference, and mechanical properties of abdominopelvic tissues: a case series. Physiother Theory Pract. 2023 Jan;39(1):49-60. doi: 10.1080/09593985.2021.2004630. Epub 2021 Nov 15. PMID 34779692
- [Background] Navarro Brazalez B, Sanchez Sanchez B, Prieto Gomez V, De La Villa Polo P, McLean L, Torres Lacomba M. Pelvic floor and abdominal muscle responses during hypopressive exercises in women with pelvic floor dysfunction. Neurourol Urodyn. 2020 Feb;39(2):793-803. doi: 10.1002/nau.24284. Epub 2020 Jan 27. PMID 31985114
- [Background] Gluppe SB, Ellstrom Engh M, Bo K. Curl-up exercises improve abdominal muscle strength without worsening inter-recti distance in women with diastasis recti abdominis postpartum: a randomised controlled trial. J Physiother. 2023 Jul;69(3):160-167. doi: 10.1016/j.jphys.2023.05.017. Epub 2023 Jun 5. PMID 37286390
- [Background] Lee N, Bae YH, Fong SSM, Lee WH. Effects of Pilates on inter-recti distance, thickness of rectus abdominis, waist circumference and abdominal muscle endurance in primiparous women. BMC Womens Health. 2023 Nov 27;23(1):626. doi: 10.1186/s12905-023-02775-5. PMID 38008749